CLINICAL TRIAL: NCT06095947
Title: The Shandong Provincial Center for Disease Control and Prevention, China
Brief Title: Exploration on the Quadrivalent Influenza Vaccine Immunization Schedule for Children Aged 3-8 Years
Status: Completed | Type: Observational
Sponsor: Hualan Biological Bacterin Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: HL-SJLG-2021-Ⅳ-02
Record Dates: First submitted 2023-09-25; First posted 2023-10-23 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: GCP
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Approximately 3ml of blood was collected on day 0, day 30 (before the second dose of inoculation), and day 60
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- There was an immunological history group: l Children who have received two or more doses of influenza vaccine (4 weeks apart) before the influenza season (2 doses of influenza vaccine do not need to be administered in the same epidemic season or consecutive epidemic season, and can be interpreted as children who have received two or more cumulative doses).
  Interventions: Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent
- There was no immunological history group: l Children who have not received or previously received <2 doses of influenza vaccine before the epidemic season.
  Interventions: Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent

INTERVENTIONS:
Biological: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent — A total of 652326 healthy children with immunization history and no immunization history aged 3-8 years who met the program requirements received two doses of normally commercially available quadrivalent influenza vaccine according to the 0,30-day procedure.

SUMMARY:
The goal of this [To evaluate the immunogenicity and safety of 1 - and 2-dose schedules of quadrivalent influenza vaccine (split virion) in healthy people with and without immunization history.] is to [aged 3-8 years] in [Healthy people]. The main question[s] it aims to answer are: • [To evaluate the immunogenicity of a two-dose schedule of quadrivalent influenza vaccine (quadrivalent influenza vaccine) in healthy population aged 3-8 years with or without vaccination history.]

•[ To evaluate whether antibody levels are different 30 days after one dose of quadrivalent influenza vaccine versus two doses of quadrivalent influenza vaccine in healthy people aged 3-8 years with or without vaccination history.]

DETAILED DESCRIPTION:
An open clinical trial design was used. A total of 652 healthy children aged 3-8 years, 326 with vaccination history and 326 without vaccination history, were selected to receive two doses of normal commercially available quadrivalent influenza vaccine according to a 0 -, 30-day schedule.

Immunogenicity: blood samples were collected for HI antibody detection before the first dose of influenza vaccine (before immunization), 30 days after the first dose of influenza vaccine (before the second dose of influenza vaccine) and 30 days after the second dose of influenza vaccine.

Adverse events (AE) were observed 30 minutes, 0-7 days and 8-30 days after each dose of vaccination by active follow-up combined with guardian reports. Occurrence of SAEs between 31 and 180 days after the second dose of vaccine.

Criteria for evaluation of immunogenicity According to the European Union seasonal influenza evaluation criteria, if the HI antibody seroconversion rate of each subtype of influenza virus was ≥40%, the HI antibody positive rate was ≥70%, and the GMI of each subtype of influenza virus was ≥2.5 times 30 days after any dose of vaccination, the vaccination schedule was considered to have acceptable immunogenicity.

Safety outcome MEASURES The occurrence of adverse reactions/events after each dose of vaccination was observed. The incidence of ① total adverse reactions/events, ② incidence of grade 3 or above adverse reactions/events and SAE, ③ incidence of adverse reactions/events severity classification, ④ incidence of adverse reactions/events by type (inoculation site and systemic, SOC, PT) and incidence of adverse reactions/events severity classification were calculated.

Note: Known adverse effects of quadrivalent influenza vaccine that have been identified in previous clinical studies are as follows:

Inoculation site (local) adverse events: pain, induration, swelling, rash, redness, pruritus, cellulitis.

Adverse events at non-inoculated sites (systemic) included fever, diarrhea, constipation, dysphagia, anorexia, vomiting, nausea, myalgia (non-inoculated sites), arthralgia, headache, cough, dyspnea, pruritus at non-inoculated sites (without skin lesions), mucocutaneous abnormalities, irritation/inhibition, acute anaphylaxis, and fatigue/fatigue.

ELIGIBILITY:
Inclusion Criteria:

* 3-8 years old;
* The legal guardian / authorized agent gives the informed consent and voluntarily signs the informed consent to comply with the requirements of the clinical trial protocol;
* Medical history, physical examination and clinical diagnosis, who to the immunization of this product.
* children who have received two or more doses of influenza vaccine (4 weeks apart) before the season of this influenza epidemic (2 doses of influenza vaccine do not need to be vaccinated in the same epidemic season or consecutive epidemic season, but can be interpreted as children who have received two or more cumulative shots).

History of l No immunization: children who had not been vaccinated or had previously received <2 doses of influenza vaccine before the influenza season.

Exclusion Criteria:

1.1.1The exclusion criteria for the first needle To l allergic to any component of the quadrialent influenza vaccine (history of any previous vaccine allergy), especially those allergic to eggs; The l axillary body temperature was 37.5℃ before inoculation;

* Any influenza vaccine (registered or research) within 6 months prior to enrollment; or planned for use during the study period;
* Use of immunoglobulin and / or any blood products within 3 months prior to enrollment; or planned for use during the study (before blood sampling);
* Patients with a history of Guillain-Barre syndrome; l Acute disease, severe chronic disease, acute onset of chronic disease, cold;
* Uncontrolled epilepsy;
* Has been diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, or other autoimmune diseases;
* those receiving immune booster or inhibitor treatment within 3 months (continuous oral or drip for more than 14 days);
* History of abnormal coagulation function (such as lack of coagulation factors, coagulation disease);
* Primary and secondary impaired immunity (history of thyroid, pancreas, liver and spleen resection);
* A history of severe allergic reactions to vaccination;
* live attenuated vaccine within 14 days before vaccination and other vaccines within 7 days before vaccination;
* Is in or recently planning to participate in other clinical trials;
* Other conditions judged by the investigator as not suitable for participation in this clinical trial.

1.1.2 Exclusion criteria for the second needle

* Patients with severe allergic reactions after the previous dose of vaccination;
* Serious adverse reactions with a causal relationship with the previous dose of vaccination; l For newly detected or those who do not meet the inclusion criteria of the first injection or meet the exclusion criteria of the first injection, the investigator will determine whether to continue to participate in the study;
* Other reasons for exclusion as considered by the investigator.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy people aged 3-8 years old
Sampling Method: Probability Sample
Enrollment: 652 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
evaluate the immunogenicity of 1-dose and 2-dose schedule in 3-8 years old healthy people with and without immunization history | Blood samples were collected before immunization, 30 days after the first dose (before the second dose) and 30 days after the first dose for influenza virus HI antibodies.
  The lower limit of the 95% confidence interval (CI) of the seroconversion rate (SCR) of hemagglutination inhibition (HAI) antibodies against each virus strain after vaccination was ≥40%. The lowest dilution used in the assay was 1 in 10. Seroconversion was defined as a prevaccination HAI titer of <1:10 and a postvaccination titer of ≥1:40 or a prevaccination titer of ≥1:10 and a 4-fold or greater increase in titer after vaccination.
evaluate the safety of one dose and two doses schedule in children aged 3-8 years | The safety was observed until 6 months after the full course of immunization
  The occurrence of adverse reactions/events after each dose of vaccination was observed. The incidence of ① total adverse reactions/events, ② incidence of grade 3 or above adverse reactions/events and SAE, ③ incidence of adverse reactions/events severity classification, ④ incidence of adverse reactions/events by type (inoculation site and systemic, SOC, PT) and incidence of adverse reactions/events severity classification were calculated.

SECONDARY OUTCOMES:
Differences in antibody levels 30 days after one dose and two doses of quadrivalent influenza vaccine among healthy people aged 3-8 years with or without vaccination history. | Blood samples were collected before immunization, 30 days after the first dose (before the second dose) and 30 days after the first dose for influenza virus HI antibodies.
  Seroconversion rate, positive rate, GMT and GMI of HI antibody against each subtype of influenza virus were calculated 30 days after the first dose and 30 days after the second dose in the vaccination history group and non-vaccination history group, respectively. The Clopper-Pearson exact probability method was used to calculate confidence intervals for rates.

CONTACTS AND LOCATIONS:
Locations (1):
- Kou Zengqiang, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided